CLINICAL TRIAL: NCT06379542
Title: Double-blind Placebo-controlled Multicenter Randomized Clinical Trial to Evaluate the Efficacy and Safety of XC8, Film-coated Tablets (Valenta Pharm JSC, Russia), in Children Aged 6-17 Years With Dry Non-productive Cough Against the Background of Acute Respiratory Viral Infection
Brief Title: Efficacy and Safety of XC8, Film-coated Tablets, in Children With Acute Respiratory Viral Infections
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XC8-03-05-2023
Record Dates: First submitted 2024-03-11; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Acute Respiratory Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XC8, film-coated tablets, 20 mg, 40 mg (Experimental): 6-12 years old: 20 mg tablet, 2 per day for 7-14 days on top of standard therapy.
  13-17 years old: 40 mg tablet, 2 per day for 7-14 days on top of standard therapy.
  Interventions: Drug: XC8
- Placebo (Placebo Comparator): 2 tablets per day for 7-14 days on top of standard therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC8 — 40 mg/day or 80 mg/day for 7-14 days
  Arms: XC8, film-coated tablets, 20 mg, 40 mg
Drug: Placebo — 2 tablets/day for 7-14 days
  Arms: Placebo

SUMMARY:
The study is planned to evaluate the therapeutic efficacy and safety of XC8, film-coated tablets, in the treatment of dry non-productive cough on the background of acute respiratory infections in children from 6 to 17 years compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patient signing the Informed Consent Form and parent/adoptive parent signing the Parent/Adoptive Informed Consent Form.
2. Male and female children between the ages of 6 and 17 years 10 months inclusive at the time of screening.
3. Clinical diagnosis of acute respiratory viral upper respiratory tract infection (J00-J06 according to ICD-10) or acute bronchitis (J20, J21 according to ICD-10).
4. Onset of disease symptoms no more than 3 days prior to screening.
5. Presence of dry non-productive cough in the patient.
6. Frequency of cough attacks ≥10 in the last 24 h before the screening visit and randomization.
7. Cough frequency rated by the patient (for patients 13-17 years of age) or parent/adoptive parent (for patients 6-12 years of age) as 3-4 points on the "daytime cough" section and 2-4 points on the "nighttime cough" Daytime and nighttime cough scales.
8. Patient (for patients 13-17 years of age) or parent/adoptive parent (for patients 6-12 years of age) assessment of cough severity on the digital rating scale as ≥4 points.
9. No indication for therapy due to BHSA infection at the time of inclusion in the study: negative rapid test for group A β-hemolytic streptococcus.
10. For patients 14-17 years of age inclusive, consent to use reliable contraceptive methods throughout study participation and for 3 weeks after the end of the study.

Reliable contraceptive methods are: sexual rest, condom use in combination with spermicide.

Non-inclusion Criteria:

1. Known or suspected hypersensitivity to the active substance or any of the excipients of the study drug/placebo.
2. Known or suspected hypersensitivity to acetylcysteine.
3. Lactose intolerance, lactase deficiency, glucose-galactose malabsorption.
4. Trauma (including open wounds in the oral cavity and erosive desquamous lesions of the oral mucosa) and/or burns of the oropharynx, scarlet fever, rubella, measles, epidemic mumps at the time of screening or within 3 months before screening.
5. Acute obstructive laryngitis or suspected obstructive laryngitis.
6. Presence of signs of laryngeal stenosis (stridor, dyspnea).
7. Exacerbation of chronic bronchitis.
8. Bronchial asthma, including history.
9. Tuberculosis in the anamnesis.
10. Emphysema of the lungs in the anamnesis.
11. Acute or chronic pneumonia or suspected pneumonia.
12. Condition after intubation.
13. Gastroesophageal reflux being the primary cause of cough (in the opinion of the investigating physician).
14. Allergic rhinitis being the primary cause of cough (in the opinion of the physician-researcher).
15. Body temperature > 39.0 °C.
16. Positive laboratory test result for SARS-CoV-2 antigen using an immunochromatographic assay at the time of screening1.
17. Need for systemic antibiotic therapy and/or other drugs/procedures on the prohibited therapy/procedure list.
18. Use of analgesics or antipyretics within 12 h prior to screening.
19. Use of glucocorticosteroids, β-adrenoblockers, ACE inhibitors, theophylline preparations, expectorants, cough suppressants, anesthetics, anti-allergic drugs (leukotriene receptor antagonists, H1-histamine receptor blockers, sodium cromoglycate preparations), antiviral drugs, immunosuppressants, systemic antibacterial agents within 7 days before screening.
20. A history of smoking.
21. History of renal or hepatic impairment.
22. History of oncologic diseases.
23. Serious cardiovascular disease at the time of screening or within 12 months prior to screening, including: severe arrhythmias requiring treatment with antiarrhythmic drugs, unstable angina pectoris, heart and coronary artery surgery, stroke.
24. Other severe, decompensated or unstable somatic diseases (any disease or condition that threatens the patient's life or worsens the patient's prognosis and makes it impossible for the patient to participate in the clinical trial).
25. Unwillingness or inability of the patient/parent/adoptive parent to comply with the protocol procedures (in the opinion of the investigating physician).
26. Pregnancy or breastfeeding period (for female patients).
27. Alcoholism, drug dependence, substance abuse history and/or at the time of screening.
28. A history of schizophrenia, schizoaffective disorder, bipolar disorder, or other psychiatric pathology.
29. Participation in another clinical trial within 3 months prior to inclusion in the study.
30. Other conditions that, in the opinion of the investigating physician, preclude the patient's inclusion in the study.

Exclusion criteria:

1. Identification of a confirmed case of COVID-19.
2. Ineffectiveness of therapy - persistence or increase in cough attack frequency ≥1 by Visit 3 (Day 8-9) compared to Visit 1 (Day 1).
3. Adverse events (AEs) requiring withdrawal of study drug/placebo.
4. Occurrence of any disease or condition during the study that, in the opinion of the investigator, worsens the patient's prognosis and makes it impossible for the patient to continue participating in the clinical trial.
5. Erroneous inclusion of a patient who does not meet the inclusion criteria and/or meets the criteria for non-inclusion.
6. Taking any of the drugs of prohibited therapy, performing a prohibited procedure.
7. Need to prescribe a prohibited concomitant therapy/procedure.
8. Pregnancy of the patient.
9. Willingness of the patient and/or his/her parent/adoptive parent to terminate the patient's participation in the study.
10. Lack of adequate cooperation of the patient and/or his/her parent/adoptive parent with the physician-researcher during the research process.
11. Other protocol violations that in the opinion of the physician-researcher are significant.
12. Other administrative reasons.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 252 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Decrease in percentage of patients with ≥50% reduction in number of cough attacs by day 5 relative to day 1 | Assessment will include data collected within 24 hours before day 1 and day 5
  Difference between the percentage of patients with ≥50% reduction in number of cough attacs by day 5 and by day 1

SECONDARY OUTCOMES:
Number of cough attacks by day 5, day 8, day 11 and day 15 | The estimate will include data collected within 24 hours before day 5, day 8, day 11 and day 15, respectively
  Number of cough attacks registered by days 5, 8, 11, and 15
Time (days) from visit 1 until clinical cough cure is achieved | The assessment will include the time from visit 1 to the first day of consecutive days on which ≤ 1 score on the "daytime cough" and "nighttime cough" sections of the scales is recorded through the end of treatment (within timeframe from 7 to 14 days)
  Clinical cure of cough is defined as having ≤ 1 score on the "daytime cough" and "nighttime cough" sections of the Daytime and Nighttime Cough Scale (a scale with scores from 0 to 5, where 0 is the absence of cough, and 5 is a severe cough that makes daytime activity impossible or a cough that makes it impossible to sleep) for at least 3 consecutive days.
Proportion of patients with presence of ≤ 1 score for the "daytime cough" and "nighttime cough" sections Daytime and nighttime cough scales by days 5, 8, 11, and 15 after visit 1 | The score for the "daytime cough" section will include data for days 4, 7, 10, and 14, respectively. The score for the "night cough" section will include data from the night prior to days 5, 8, 11, and 15, respectively.
  Score on the "daytime cough" and "nighttime cough" sections of the Daytime and Nighttime Cough Scale (a scale with scores from 0 to 5, where 0 is the absence of cough, and 5 is a severe cough that makes daytime activity impossible or a cough that makes it impossible to sleep)
Change (score) in cough severity by digital rating scale by days 5, 8, 11 and 15 compared to visit 1 | The score will include data 24 h before days 5, 8, 11 and 15, respectively
  Score assessed with digital rating scale (a scale from 0 to 10, where 0 is the absence of cough, and 10 is the most excruciating cough imaginable)
Percentage of patients needed acetylcysteine | Day 1 - Day 21±2
  Percentage of patients who were prescribed a preparation with acetylcysteine for transition of dry cough to wet cough
Proportion of patients with complete resolution of all symptoms of acute respiratory infection by days 4, 7, 10 and 14 | Days 4, 7, 10, 14
  Complete resolution of all symptoms is defined as achieving a score of 0 for each symptom on the Basic Symptom Rating Scale for acute respiratory infections (a 6-item inventory including Fatigue, Sore throat, Nasal congestion, Rhinorrhea, Myalgia, and Headache, assessed using a score from 0 to 3, where 0 is the absence of the symptom, and 3 is the most severe symptom severity)
Percentage of patients with each category of Global Physician-Researcher Assessment of Therapy Effectiveness at visits 2, 3, 4, and 5 | Day 3-16
  Assessment of clinical effectiveness using Global Physician-Researcher Assessment of Therapy Effectiveness (a 5-point scale, where 1 is the absence of efficacy, and 5 is very high efficiency, meaning a complete cure of coughs)
Number of adverse events (AEs) | Day 0 - Day 21±2
  Total number of AEs stratified by severity and frequency
Adverse reactions | Day 0 - Day 21±2
  Frequency of adverse reactions
Serious adverse events (SAEs) | Day 0 - Day 21±2
  Frequency of serious adverse events (SAEs) associated with study drug/placebo use
Percentage of patients with AEs | Day 0 - Day 21±2
  Percentage of patients with at least one AE
Percentage of patients who interrupted treatment | Day 0 - Day 21±2
  Percentage of patients who interrupted treatment due to AE

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - City Pediatric Outpatient Clinic number 5, Perm
  - Professors' Clinic LLC., Perm
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 44", Saint Petersburg
  - ArsVite North-West, LLC, Saint Petersburg
  - PiterKlinika LLC, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Pediatric Polyclinic No. 35", Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided